CLINICAL TRIAL: NCT00542854
Title: A Pilot Study on the Effects of Digital Music Players on Implantable Cardioverter Defibrillators and Pacemakers in Pediatrics and Congenital Heart Disease
Brief Title: iPod and Other MP3 Players on ICDs and Pacemakers in Children
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Charles Berul, MD - Principal Investigator, Children's Hospital Cardiology
Other Study IDs: CHB-07-08-0308
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Heart Block; Bradycardia; Tachycardia; Arrhythmia
Keywords: arrhythmia; pacemaker; defibrillator; electromagnetic interference
MeSH Terms: conditions — Heart Block; Bradycardia; Tachycardia; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MP3: 4 different brands of MP3 players will be tested at 3 distances from pacemakers and ICDs.
  Interventions: Device: MP3

INTERVENTIONS:
Device: MP3 — 4 different brands of MP3 players will be tested at 3 distances from ICD/pacemaker site in children and adults with congenital heart disease.

SUMMARY:
Unlike phones, which are commonly held to the ear, music is now available via portable MP3 players and they can be held almost anywhere. Thaker et al state that Apple iPods cause pacemaker interference in 50% of their patients, with over-sensing in 20% of patients, telemetry interference in 29% of patients and pacemaker inhibition in 1.2% of patients. The mean age for their sample was 76.1 years +/- 8.6 years. We anticipate that a higher proportion of teenagers and children who have pacemakers use portable MP3 players than in the elderly adult population.We will include the first 100 patients with pacemakers and ICDs who consent for the prospective observational study a single tertiary care center. We intend to conduct a descriptive study, tabulating the number of times that a pacemaker or ICD has changes in the sensing thresholds, pacing thresholds, telemetry interference or pacemaker inhibition when exposed to a series of portable MP3 players at various distances. In addition, we will describe the nature and quantitative differences of those changes.

DETAILED DESCRIPTION:
Since pacemakers and implantable cardioverter defibrillators (ICDs) have been used, there have been questions about what external sources interference could alter their functioning or event recording properties. Because these devices are often intended to be life-saving, their proper functioning is of critical importance.

The literature documents a number of common sources of possible interference. Interference with MRI and electrocautery have been observed (1, 2). Outside the hospital, store security devices and personal digital assistants (PDAs) have been evaluated (3, 4). In 1997, Hayes et al published a randomized, prospective trial concluding that cellular telephones impacted the functioning of pacemakers, but that they did not seem to have any effect at any significant distance (5). They showed that a phone being used at the ear was sufficiently far away to prevent a health risk and recommended that phones not be put in shirt pockets or used near the device.

Unlike phones, which are commonly held to the ear, music is now available via portable MP3 players and they can be held almost anywhere. Thaker et al state that Apple iPods cause pacemaker interference in 50% of their patients, with over-sensing in 20% of patients, telemetry interference in 29% of patients and pacemaker inhibition in 1.2% of patients (6). The mean age for their sample was 76.1 years +/- 8.6 years. We anticipate that a higher proportion of teenagers and kids who have pacemakers use portable MP3 players than in the elderly adult population.

Design Prospective observational study a single tertiary care center.

Subjects

The electrophysiology department at Children's Hospital, Boston follows a large number of patients with pacemakers and ICDs. Approximately 15 patients are seen each week in clinic for routine pacemaker evaluation.

Entry Criteria We will include the first 100 patients with pacemakers and ICDs who consent for the prospective trial.

1. Consent for participation
2. Active pacemaker/ICD, which is functioning appropriately at the time of interrogation based on internal diagnostics and the judgment of an appropriate clinician (electrophysiology nurse, fellow and/or attending.
3. Normally functioning leads and thresholds at the time of interrogation based on internal diagnostics and the judgment of an appropriate clinician (electrophysiology nurse, fellow and/or attending.

Variables

Primary Outcome Change in pacemaker sensing thresholds, pacing thresholds, telemetry interference or pacemaker inhibition.

Methods

Study investigators will first obtain informed consent from each patient or family and, where appropriate, assent from the child.

At the conclusion of their routine clinic visit, each patient will have his or her pacemaker attached to the appropriate proprietary interrogation system for their pacemaker device. We will then monitor the pacemaker/ICD system while placing a series of portable music devices at various distances from the pacemaker/ICD system: (1) 2cm, (2) 30cm, (3) 100cm. At each distance the pacemaker will be re-interrogated for changes in pacemaker sensing thresholds, pacing thresholds, telemetry interference or pacemaker inhibition. At the end of the testing process, the devices will be removed from near the patient and the device will be interrogated again to assure that the device is at the appropriate clinical settings.

Risks

We believe that there are no more than minimal risks associated with this study. The principle intervention is the placement of a music device near the pacemaker/ICD during the time of pacemaker monitoring. We consider this risk to be similar to the risks encountered by many patients who are currently using portable music devices outside the hospital. In addition, we do not expect any permanent change in the pacemaker or ICD settings, thresholds or functioning.

Statistical Issues

Hypothesis Our hypothesis is that the close approximation of portable MP3 players interfere with the appropriate sensing and recording of pacemakers and ICDs.

Sample Size and Power Calculations We intend to conduct a descriptive study, tabulating the number of times that a pacemaker or ICD has changes in the sensing thresholds, pacing thresholds, telemetry interference or pacemaker inhibition when exposed to a series of portable MP3 players at various distances. In addition, we will describe the nature and quantitative differences of those changes.

Because we do not intend to do comparisons for significance against a control group, we have chosen 100 patients as a reasonable sample size for evaluating possible changes in pacemaker/ICD function.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults with congenital heart disease who have an implanted pacemaker or defibrillator

Exclusion Criteria:

* Age less than 4 or inability to communicate adequately with study team

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adults with congenital heart disease who have an implanted pacemaker or defibrillator
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in pacemaker sensing thresholds, pacing thresholds, telemetry interference or pacemaker inhibition. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Charles Berul, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States